CLINICAL TRIAL: NCT02468505
Title: STEPS: Stepped Transition in Education Program for Students With ASD
Acronym: STEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Yasuo Miyazaki, Associate Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R34MH104337 (NIH)
Record Dates: First submitted 2015-06-04; First posted 2015-06-11 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Structured transition support program; Transition 'as usual'
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STEPS (Experimental): structured psychosocial transition support that includes individual counseling, and education/training for parent and school personnel
  Interventions: Behavioral: STEPS
- TAU (No Intervention): typical transition services and supports

INTERVENTIONS:
Behavioral: STEPS — time-limited behavioral counseling, online materials, training
  Arms: STEPS

SUMMARY:
Young adults who have Autism Spectrum Disorder (ASD) without co-occurring intellectual impairment face a fairly unique set of challenges as they transition out of secondary school. These students are often quite capable of succeeding in higher education and many of them have interest in pursuing advanced degrees, but the nature of their disability and associated deficits (e.g., poor time management and poor self-regulation) may impede success. Individualized, appropriately timed, and developmentally sensitive transition and support services may promote optimal outcomes for these young people. The goal of this project is to develop a comprehensive program to promote successful transition of students with ASD from high school to post-secondary education.

DETAILED DESCRIPTION:
The investigators propose to refine and then evaluate a novel transition support and intervention program for adolescents and young adults with ASD: STEPS [Stepped Transition in Education Program for Students with ASD]. By targeting improved self-regulation (SR) and self-determination (SD) in young people with ASD, the investigators assert that this program may have positive outcomes with respective to college adjustment and functional behavior. Although the program will be finalized during the first phase of the proposed project, at present STEPS is comprised of two levels (or steps), which match the student's particular needs in relation to transition planning. In Step 1, students facing transition (i.e., have identified the college they will attend (either 2-year or 4-year institution) but are still in high school) and their caregivers will receive information to assist in transition planning, undergo readiness self-assessments (to identify degree of preparedness for post-secondary school), and participate in interactive sessions online and in person to promote self-knowledge and determination. The goal of Step 1 is to assist families and students with transition planning, specifically ensuring that families and students have the tools needed to make informed choices and take necessary steps (e.g., remediating identified skill deficits) to increase the likelihood of a successful transition out of high school. In Step 2, college students with ASD will receive fairly intensive supports and interventions, including individual counseling, structured support services, social integration activities, and coaching to promote academic and social success. The following specific aims are proposed.

ELIGIBILITY:
Inclusion Criteria:

* Must be 16 to 25 years
* Must have clinical diagnosis of autism spectrum disorder
* Must be preparing for postsecondary education or enrolled in postsecondary education

Exclusion Criteria:

* Intellectual disability
* Psychiatric disturbance that warrants immediate treatment

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2018-07-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure feasibility and program acceptability | 16 weeks
  parent- and youth self-report measure of utility of program, acceptability, and consumer satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Polytechnic Institute and State University, Blacksburg, Virginia, United States